CLINICAL TRIAL: NCT06221280
Title: Effects of Transversus Abdominis and Erector Spina Plane Blocks on Post-Cesarean Pain Control and Postpartum Depression
Brief Title: Effects of Nerve Blocks on Pain After Caesarean Section and Postpartum Depression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Feyza Calisir, Assistant professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/10-02
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain; Cesarean Section; Postpartum Depression
Keywords: Nerve block, cesarean, postpartum depression
MeSH Terms: conditions — Pain, Postoperative; Depression, Postpartum | interventions — Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group E (Active Comparator): Patients who underwent erector spinae plane block
  Interventions: Procedure: Nerve block
- Group T (Active Comparator): Patients who underwent transversus abdominis plane block
  Interventions: Procedure: Nerve block

INTERVENTIONS:
Procedure: Nerve block — Group E: While performing the erector spina plan block; Patients are placed in the lateral decubitus position, aseptic conditions are provided, the spinous process in the midline is determined under ultrasonography guidance, and the transverse process is determined 3 cm laterally from the T11 level. 100 mm 22G block needle erector.
  Group T: The lumbar petit region will be determined and placed on the lateral abdominal wall at the mid-axillary line, between the iliac crest and the lower costal arch, via a linear probe (12-15 MHz probe). After determining the internal oblique muscle as the thickest muscle and the transversus abdominis muscle as the thinnest muscle, a 100 mm 22 G needle will be placed in the same plane as the USG probe (in-plane or long axis technique). The progress of the needle will be observed on ultrasound along with the facial click sensation. After the second click sensation is felt between the internal oblique and transversalis fascia.

SUMMARY:
At the end of your cesarean section surgery, which is started by applying medication to the spinal cavity from your waist, pain medication will be applied between the relevant muscle and its covering from your lower abdomen or back with the help of ultrasonography and a special block needle. Then, a patient-controlled pain device with a serum containing painkillers will be connected to your vascular access, and its use and purpose will be explained to you. You will be asked about your pain condition and the severity score of your pain, if any, at certain hourly intervals. At the end of 24 hours, a pain device will be removed, your satisfaction will be questioned and your complaints, if any, will be recorded. Immediately before surgery and 4-6 days after your surgery. An evaluation survey consisting of 10 questions will be asked to you within a 5-minute period during the weeks, at a time when you are free, and your answers will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Having a good mental status,
2. Those aged ≥18 years,
3. Term pregnant (gestational age ≥ 36 weeks),
4. American Society of Anesthesiologists class II-III,
5. Patients who underwent cesarean section with spinal anesthesia will be included.

Exclusion Criteria:

1. Having labor at term or obstetric emergency,
2. Having a twin pregnancy,
3. Having a diagnosed psychiatric disorder/using psychiatric medication,
4. Those who are allergic to local anesthetics and/or drugs used in the study,
5. The patient-controlled anesthesia device is out of use for any reason within the first 24 hours postoperatively,
6. Having peripheral neuropathy or neuromuscular disease,
7. Patients using anticoagulant drugs that will prevent regional anesthesia will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Application in cesarean section cases
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS score) | 12 months
  Evaluation of the postoperative analgesic effectiveness of erector spinae and transversus abdominis plane blocks after cesarean section

SECONDARY OUTCOMES:
Postpartum depression (Edinnburg Depression Scale) | 12 months
  Comparison of the effectiveness of blocks for analgesia in terms of postpartum depression

CONTACTS AND LOCATIONS:
Locations (1):
- KahramanmarasSIU, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)